CLINICAL TRIAL: NCT03719040
Title: Physiologic Pacing Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10270
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Bradycardia; Sinus Node Dysfunction; Heart Block; Syncope; Cardiomyopathies; Ventricular Tachycardia; Heart Failure
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Heart Block; Syncope; Cardiomyopathies; Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Physiologic pacing device implant — An alternative and potentially more effective pacing strategy for patients with electrical conduction abnormalities is physiologic pacing. Physiologic pacing is achieved by delivering a pacing stimulus to a cardiac conduction structure, such as the bundle of His or left bundle branch (LBB) of the His-Purkinje system, with a permanent lead. Physiologic pacing activates the heart through the native His-Purkinje conduction system, thus offering the most physiologic pacing approach to correct electrical dyssynchrony. Physiologic pacing has emerged as a feasible and safe alternative to pacemaker therapy and CRT with clinical and electrophysiological advantages.

SUMMARY:
The Physiologic Pacing Registry is a prospective, observational, multi-center registry performed to gain a broader understanding of 1) physiologic pacing implant and follow-up workflows, including pacing and sensing measurements and 2) the clinical utility in creating a 3-dimensional electro-anatomical map of cardiac structures prior to physiologic pacing device implants based on the clinical site's routine care.

DETAILED DESCRIPTION:
The Physiologic Pacing Registry will be conducted to gain a deeper understanding of physiologic pacing device implants and follow-up workflows, including device and programmer measurements to help inform Abbott's product and clinical data development efforts. Additionally, the registry will provide a broader understanding of the clinical utility in mapping physiologic pacing structures with the use of Abbott's EnSite Cardiac Mapping System with an electrophysiology catheter prior to device implants for those institutions where mapping is routine care prior to physiologic pacing device implant.

The registry will include patients undergoing implantation of an Abbott pacemaker, defibrillator, or a cardiac resynchronization therapy (CRT) pacemaker (CRT-P) or CRT defibrillator (CRT-D) according to the clinical site's routine care. Only patients scheduled to receive an Abbott device may be enrolled to ensure proper device data collection for future software and other physiologic pacing product development. The decision to provide physiologic pacing therapy and selection of devices for implant are at the discretion of the implanting physician. Abbott will collect data on the use of all commercially available leads and associated implant tools based on the physician's discretion as part of routine clinical practice within the registry.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for implantation of an Abbott pacemaker, defibrillator, or CRT-P/D device with any commercially available pacing lead as part of a physiologic pacing procedure according to the clinical site's routine care.
2. At least 18 years of age.
3. Willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
4. Provided written informed consent prior to any registry-related procedures.

Exclusion Criteria:

1. History of tricuspid valve repair or replacement.
2. Currently participating in another clinical study with an active treatment arm and belong to the active arm
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the registry or to comply with follow-up requirements, or impact the scientific soundness of the registry results.
4. Chronic physiologic pacing lead implanted
5. Life expectancy of < 6 months.
6. Known contraindication for physiologic pacing therapy/implant (i.e. ongoing infection, known occlusion of the subclavian vein, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The registry will include patients undergoing implantation of a pacemaker, defibrillator, or a cardiac resynchronization therapy (CRT) pacemaker (CRT-P) or CRT defibrillator (CRT-D) according to the clinical site's routine care.
Sampling Method: Non-Probability Sample
Enrollment: 870 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwangdeok Lee, Study Director — Abbott
Locations (50):
- United States (26):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Mills-Peninsula Medical Center, Burlingame, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Yoel R. Vivas, MD, Delray Beach, Florida
  - Usman R. Siddiqui, MD, Winter Park, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - IU Health Bloomington Hospital, Bloomington, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Providence Hospital, Southfield, Michigan
  - The Valley Hospital, Ridgewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New York University Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Texas Cardiac Arrhythmia, Austin, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - St. Joseph Medical Center, Tacoma, Washington
- Australia (3):
  - The Northern Hospital, Epping, Victoria
  - Mulgrave Private Hospital, Mulgrave, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Universitätsklinik Graz, Graz, Styria, Austria
- Canada (2):
  - QE II Health Sciences, Halifax, Nova Scotia
  - CHUS Fleurimont, Sherbrooke, Styria
- Fakultni nemocnice Kralovske Vinohrady, Prague, Central Bohemia, Czechia
- France (2):
  - CHRU Rouen Hospital Charles Nicolle, Rouen, Upper Normandy
  - Clinique Ambroise Pare, Neuilly-sur-Seine, Île-de-France Region
- Germany (2):
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
- Prince of Wales Hospital, Hong Kong, Hong Kong SAR, Hong Kong
- India (2):
  - Fortis Memorial Research Institute, Gurugramam, Haryana
  - Asian Institute of Gastroenterology (AIG) Hospital, Hyderabad
- Italy (2):
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Ospedale S.Maria della Misericordia, Rovigo
- Maastricht University Medical Center, Maastricht, Netherlands
- Gornoslaskie Centrum Medyczne im.prof. Leszka Gieca, Katowice, Poland
- Singapore (2):
  - National Heart Centre Singapore, Singapore, Central
  - NG Teng Fong General Hospital, Singapore, Central
- Christiaan Barnard Memorial Hospital, Cape Town, South Africa
- Spain (2):
  - Hospital Universitario Virgen de la Nieves, Granada
  - Hospital General Juan Ramon Jimenez, Huelva
- Center Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vazquez PM, Mohamed U, Zanon F, Lustgarten DL, Atwater B, Whinnett ZI, Curila K, Dinerman J, Molina-Lerma M, Wiley J, Grammatico A, Lee K, Vijayaraman P. Result of the Physiologic Pacing Registry, an international multicenter prospective observational study of conduction system pacing. Heart Rhythm. 2023 Dec;20(12):1617-1625. doi: 10.1016/j.hrthm.2023.06.006. Epub 2023 Jun 20. PMID 37348800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 870 subjects were enrolled in the registry
Groups:
- Physiologic Pacing Registry: The registry is a prospective, single arm, observational, multi-center study to gain a broader understanding of physiologic pacing implant and follow-up workflows, including pacing and sensing measurements. Subjects scheduled for implantation of an Abbott pacemaker, defibrillator, or CRT-P/D device with any commercially available pacing lead as part of a physiologic pacing procedure according to the clinical site's routine care were enrolled in the registry.
Period: Overall Study
Arm/Group | Physiologic Pacing Registry
Started | 870
Attempted Implant | 849
1-Month Follow up | 731
6-Month Follow up | 667
Completed | 667
Not Completed | 203
Not completed — Withdrawal by Subject | 177
Not completed — Lost to Follow-up | 26

BASELINE CHARACTERISTICS:
Population: The patient population for this registry was potential subjects undergoing implantation of an Abbott pacemaker, defibrillator, or CRT-P/D with any market released pacing lead as part of a physiologic pacing procedure according to the clinical site's routine care.
Groups:
- Physiologic Pacing Registry: The registry is a single arm study
Arm/Group | Physiologic Pacing Registry
Number analyzed (Participants) | 870
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337
  Male | 533
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135
  Not Hispanic or Latino | 702
  Unknown or Not Reported | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 789
  More than one race | 0
  Unknown or Not Reported | 17
NYHA Class [Count of Participants; unit: Participants] — Population: NYHA classification was evaluated only in 485 subjects.
  The New York Heart Association (NYHA) functional classification system categorizes congestive heart failure patients based on their symptoms and physical activity limitations. The classes used in this system are I to IV, with I indicating less severity and higher numbers indicating greater severity.
  Participants
    number analyzed (Participants) | 485
    Class I | 98
    Class II | 241
    Class III | 137
    Class IV | 9
Cardiomyopathy Type [Count of Participants; unit: Participants]
  Non-ischemic | 145
  Ischemic | 134
  Idiopathic | 5
  None | 586

OUTCOME MEASURES:

1. Primary Outcome: Physiologic Pacing Implant Success Rate
Description: 849 subjects underwent attempted implants of physiologic pacing leads. Implant success rate was based on investigator-reported outcome.
Time Frame: During procedure
Population: The patient population for this analysis includes subjects underwent implantation of an Abbott pacemaker, defibrillator, or CRT-P/D with any market released pacing lead as part of a physiologic pacing procedure according to the clinical site's routine care.
Measure: Count of Participants; unit: Participants
Arm/Group | Physiologic Pacing Registry
Number analyzed (Participants) | 849
Participants | 768

2. Primary Outcome: Pacing Capture Threshold for His Bundle Pacing
Description: The pacing capture threshold was collected to characterize electrical performance in the Bundle of His area at 6 months. Pacing capture threshold is the minimum amount of voltage (V) needed to depolarize the myocardium or heart muscle with an electrical impulse from a pacemaker, ICD, or CRT.
Time Frame: 6 Months
Population: Subjects who did have a pacing lead implant successfully in bundle of His and complete the 6-month visit.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Physiologic Pacing Registry
Number analyzed (Participants) | 420
Volts | 1.59 (0.97)

3. Post Hoc Outcome: Pacing Capture Threshold for Left Bundle Branch Area Pacing
Description: The pacing capture threshold was collected to characterize electrical performance in the Left Bundle Branch area at 6 months. Pacing capture threshold is the minimum amount of voltage (V) needed to depolarize the myocardium or heart muscle with an electrical impulse from a pacemaker, ICD, or CRT.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Physiologic Pacing Registry
Number analyzed (Participants) | 209
Volts | 0.79 (0.33)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Physiologic Pacing Registry
All-Cause Mortality (participants affected / at risk) | 23/870
Serious Adverse Events (participants affected / at risk) | 95/870
Other Adverse Events (participants affected / at risk) | 47/870
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physiologic Pacing Registry (N=870)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Exacerbation Of Heart Failure (Cardiac disorders) | 8 (11)
Atrial Fibrillation (Cardiac disorders) | 6 (6)
Atrial Extrasystole (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Nonsustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Pleural Effusion (Cardiac disorders) | 1 (1)
Premature Atrial Complex (Cardiac disorders) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 1 (1)
Rapid Atrial Flutter (Cardiac disorders) | 1 (1)
Unstable Angina (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 3 (3)
Intestinal Lesions (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 4 (4)
Decrease In General State Of Health (General disorders) | 2 (2)
Acute Respiratory Distress Syndrome (General disorders) | 1 (1)
Bed Rest Syndrome (General disorders) | 1 (1)
Cancer (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Exacerbation Of Heart Failure (General disorders) | 1 (1)
Falls (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Infection (General disorders) | 1 (1)
Multiorgan Failure (General disorders) | 1 (1)
Cholecystolithiasis (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 17 (19)
Covid 19 Infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Fever Of Unknown Origin (Infections and infestations) | 1 (1)
Lower Leg Swelling (Infections and infestations) | 1 (1)
Pocket Erosion (Infections and infestations) | 1 (1)
Worsening Mitral Regurgitation (Infections and infestations) | 1 (1)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 3 (3)
Pneumothorax (Injury, poisoning and procedural complications) | 3 (3)
Cardiogenic Shock (Injury, poisoning and procedural complications) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Infection (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1)
Stroke (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 (1)
Twiddler's Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Atypical Fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizures (Nervous system disorders) | 1 (3)
Stroke (Nervous system disorders) | 1 (1)
Lead Migration/Dislodgement (Product Issues) | 12 (12)
Rise In Threshold/Elevated Pacing Threshold (Product Issues) | 3 (3)
Exit Block (Product Issues) | 1 (1)
Extracardiac Stimulation (Phrenic Nerve, Diaphragm, Chest Wall) (Product Issues) | 1 (1)
Lead Malfunction Due To Conductor Fracture/Lead Fracture (Product Issues) | 1 (1)
Loss Of Normal Device Function Due To Battery Failure Or Component Malfunction (Product Issues) | 1 (1)
Pocket Erosion (Product Issues) | 1 (1)
Undersensing (Product Issues) | 1 (1)
Possible Post Traumatic Stress Disorder (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pocket Erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physiologic Pacing Registry (N=870)
Complete Heart Block (Cardiac disorders) | 1 (1)
Pacemaker-Mediated Tachycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Dyspnea (General disorders) | 2 (2)
Dizziness (General disorders) | 1 (1)
Left Upper Extremity Edema (General disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Hematoma/Seroma (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Lead Migration/Dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Swelling At Incision Site And Left Arm (Injury, poisoning and procedural complications) | 1 (1)
Thromboemboli (Injury, poisoning and procedural complications) | 1 (1)
Hematoma/Seroma (Investigations) | 1 (1)
Lead Migration/Dislodgement (Product Issues) | 10 (10)
Rise In Threshold/Elevated Pacing Threshold (Product Issues) | 10 (10)
Loss Of Pacing And/Or Sensing (Product Issues) | 7 (7)
Extracardiac Stimulation (Phrenic Nerve, Diaphragm, Chest Wall) (Product Issues) | 2 (2)
Oversensing (Product Issues) | 2 (2)
Interruption Of Desired Pulse Generator Function Due To Electrical Interference (Product Issues) | 1 (1)
Lead Malfunction Due To Conductor Fracture/Lead Fracture (Product Issues) | 1 (1)
Undersensing (Product Issues) | 1 (1)
Left Upper Extremity Edema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03719040/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03719040/SAP_001.pdf